CLINICAL TRIAL: NCT04802317
Title: Identifying the Relationship Between the Features of the Composition and Functioning of the Intestinal Microbiota With the Course of Chronic Obstructive Pulmonary Disease and Asthma (MicrObAs)
Brief Title: Intestinal Microbiota in COPD and Asthma
Acronym: MicrObAs
Status: Completed | Type: Observational
Sponsor: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Collaborators: Center for Strategic Planning and Management of Biomedical Health Risks (Unknown)
Responsible Party: Sponsor
Other Study IDs: 03-08/20
Record Dates: First submitted 2021-03-12; First posted 2021-03-17 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Chronic Respiratory Diseases
Keywords: intestinal microbiota; COPD; asthma; lipopolysaccharides; trimethylamine-N-oxide; course of the diseases; exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: Health people without any respiratory diseases
  Interventions: Diagnostic Test: Identification of the composition of the intestinal microbiota
- Bronchial asthma: Patients with asthma
  Interventions: Diagnostic Test: Identification of the composition of the intestinal microbiota
- COPD: Patients with chronic obstructive pulmonary disease
  Interventions: Diagnostic Test: Identification of the composition of the intestinal microbiota

INTERVENTIONS:
Diagnostic Test: Identification of the composition of the intestinal microbiota — Identification of the composition of the intestinal microbiota

SUMMARY:
The composition of the intestinal microbiota, the level of lipopolysaccharides, TMAO in the blood, and other parameters of patients with COPD (n=50), asthma (n=50) and the control (n=40) will be assessed as factors associated with exacerbations and respiratory symptoms in the prospective study (12 months).

DETAILED DESCRIPTION:
The patients from "Biobank of blood and feces for the development of a clinical and biological platform as a basis for an innovative approach to the prevention of chronic non-infectious diseases based on the composition of the intestinal microbiota" study will be included (cross-sectional study). The protocol of the above study included the assessment of socio-demographic, anthropometric data, clinical blood pressure (BP), ECG, blood tests, fecal microbiota studies, spirometry data, diet questionnaire. ABPM, HBP, other questionnaires (mMRC, CAT, ACQ-5, GMBQ) will be added to initial data (=visit 1). Than the four visits (2-5th visits) in 3 each months will be performed to assess respiratory symptoms, exacerbations of COPD/asthma, respiratory infections, therapy, BP, and other parameters. The standard statistical methods will be used.

ELIGIBILITY:
Inclusion Criteria:

for control group:

* Normal spirometry results with bronchodilation test (salbutamol 400 mcg);
* Absence of COPD, asthma, chronic bronchitis and other lung diseases
* BMI<40kg/m2

for asthma/COPD groups:

* Primary medical documentation confirming the diagnosis of COPD or asthma
* Regular therapy for COPD, asthma and any chronic disease for at least 4 weeks prior to enrollment in this study.
* FEV1 / FVC <0.70 after inhalation of 400 mcg of salbutamol for patients with COPD
* BMI<40kg/m2

Exclusion Criteria:

* Exacerbation of chronic noninfectious diseases, including exacerbation of COPD / asthma, within 4 weeks prior to enrollment in this study.
* Exacerbation of COPD or asthma in the next 3 months, requiring the treatment of antibiotic therapy or systemic corticosteroids;
* Cerebral stroke, transient ischemic attack or myocardial infarction within 6 months before the date of enrollment in the study;
* Clinically significant chronic diseases (oncological, systemic diseases of the connective tissue, diseases of the blood system, heart failure, Crohn's disease, ulcerative colitis, etc. according to anamnesis);
* GFR <30 ml / min / 1.73m2;
* Atopy in a patient with COPD or a control group (any allergic manifestations - skin, nasal, conjunctival, food, etc.);
* Chronic respiratory diseases in a patient of the control group (COPD, asthma, chronic bronchitis, interstitial lung diseases);
* History of organ transplantation;
* Mental illness;
* Intestinal infection (food poisoning) in the next 3 months;
* Other acute infectious diseases. It is possible to turn on not earlier than 4 weeks after complete recovery and cessation of treatment;
* History of severe COVID-19;
* HIV infection, chronic viral hepatitis according to the history;
* Clinically significant oncological disease;
* Pregnancy and lactation;
* Alcoholism, taking narcotic drugs;
* Taking antimicrobial, probiotic drugs and systemic corticosteroids during the last 3 months;
* Genetic engineering / biological therapy.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients without COPD, asthma, chronic bronchitis and other lung diseases for control group. Patients asthma/COPD with for asthma/COPD groups.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Exacerbation of asthma / chronic obstructive pulmonary disease | 12 months
  Number of patients with exacerbation of bronchial asthma or chronic obstructive pulmonary disease, number of exacerbation per year

CONTACTS AND LOCATIONS:
Overall Officials: Marina Smirnova, PhD, MD, Principal Investigator — NRCPM
Locations (1):
- NRCPM, Moscow, Russia